CLINICAL TRIAL: NCT06493149
Title: Tensegrity Principle in Massage Therapy on Selected Anatomical Examples
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Wroclaw University of Health and Sport Sciences (Other)
Responsible Party: Principal Investigator, Krzysztof Kassolik, Phd, Professor, Wroclaw University of Health and Sport Sciences
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: WroclawUHSS1
Record Dates: First submitted 2024-06-26; First posted 2024-07-09 (Actual); Last update posted 2025-09-12 (Actual); Status verified 2025-09

CONDITIONS: Healthy
Keywords: Massage therapy, tensegrity
MeSH Terms: interventions — Massage

STUDY DESIGN:
Intervention Model Description: a randomised, controlled, parallel, two-arm trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Tensegrity massage group (Experimental): Participants in the tensegrity massage group are provided with the 5-minute massage session in the anterior compartment muscles of the forearm, tensor fasciae latae muscle, brachioradialis muscle, deltoid muscle, latissimus dorsi muscle and peroneus longus muscle.
  Interventions: Other: Massage therapy
- Massage group (Active Comparator): Participants in the massage group are provided with the 5-minute massage session in the anterior compartment muscles of the forearm, tensor fasciae latae muscle and brachioradialis muscle
  Interventions: Other: Massage therapy

INTERVENTIONS:
Other: Massage therapy — Participants receive a Swedish massage based on the tensegrity principle.

SUMMARY:
The study design is a randomised, controlled, parallel, two-arm trial. The subjects are randomly assigned to one of the study groups: the intervention group or the control group. The study will analyze the applicability of the tensegrity principle in the massage therapy. The main aim of this study is to examine if the tensegrity principle can be used in massage therapy to increase the effectiveness of the intervention. Contractile and passive mechanical properties are assessed before and after the intervention.

DETAILED DESCRIPTION:
The phenomenon of tensegrity, despite the ever-growing interest and its many supporters, still remains a theoretical model. Its assumptions refer to the possibility of spreading stresses between individual elements of the musculoskeletal system in order to achieve structural homeostasis. An important role here is played by muscles that remain in structural contact with each other, e.g. through a common bone attachment or fascia. Theoretically, this means that a change in the tone of one muscle can lead to changes in the tone of other muscles that are structurally connected to it. It is worth noting that this mechanism works both when one of the muscles increases its tension and when this tension is decreased.

The difficulty associated with assessing the significance of tensegration for the motion system consists in the proper design of research that accurately quantifies this phenomenon. Experiments conducted to date have mostly been performed in vitro. Despite their scientific value, analyses of this type only take part of this phenomenon into account, because they do not consider the presence of body fluids as well as the tension produced by nerves and blood vessels.

In this project the following connection between muscles are tested:

* deltoid muscle and brachioradialis muscle
* latissimus dorsi muscle and the anterior compartment muscles of the forearm,
* tensor fasciae latae and pectoralis major muscle

ELIGIBILITY:
Inclusion Criteria:

* age between 18 and 24 years;
* healthy individuals, with no lower and upper extremities pathology;
* PA≥600 MET-min/week assessed by IPAQ questionnaire;
* no medical contraindication of massage therapy;
* body mass index 18,5 < BMI ≤ 25kg/m2
* signing the informed consent.

Exclusion Criteria:

* individuals suffering from neurologic or orthopaedic problems;
* lower ot upper extremities surgical interventions;
* cancers;
* musculoskeletal disorders
* body mass index 18,5 > BMI ≥ 25kg/m2
* the lack of informed consent.

Ages: 18 Years to 24 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 80 (Estimated)
Dates: Start 2024-06-01 (Actual); Primary Completion 2024-07-20 (Actual); Study Completion 2025-10-31 (Estimated)

PRIMARY OUTCOMES:
Change in maximal displacement of the deltoid muscle after therapy compared to baseline | 1) baseline, 2) immediately after the massage session
  The maximal radial displacement is produced in the muscle belly after the electrical stimulation. Measuring device: TMG S2, Change = (Value after therapy - baseline)
Change in maximal displacement of the latissimus dorsi muscle after therapy compared to baseline | 1) baseline, 2) immediately after the massage session
  The maximal radial displacement is produced in the muscle belly after the electrical stimulation. Measuring device: TMG S2, Change = (Value after therapy - baseline)
Change in maximal displacement of the and peroneus longus muscle after therapy compared to baseline | 1) baseline, 2) immediately after the massage session
  The maximal radial displacement is produced in the muscle belly after the electrical stimulation. Measuring device: TMG S2, Change = (Value after therapy - baseline)
Change in delay time of the deltoid muscle after therapy compared to baseline. | 1) baseline, 2) immediately after the massage session
  Delay time is the time in which the muscle displacement increases to 10% after the electrical stimulation. Measuring device: TMG S2, Change = (Value after therapy - baseline)
Change in delay time of the latissimus dorsi muscle after therapy compared to baseline. | 1) baseline, 2) immediately after the massage session
  Delay time is the time in which the muscle displacement increases to 10% after the electrical stimulation. Measuring device: TMG S2, Change = (Value after therapy - baseline)
Change in delay time of the peroneus longus muscle after therapy compared to baseline. | 1) baseline, 2) immediately after the massage session
  Delay time is the time in which the muscle displacement increases to 10% after the electrical stimulation. Measuring device: TMG S2, Change = (Value after therapy - baseline)
Change in contraction time of the deltoid muscle after therapy compared to baseline. | 1) baseline, 2) immediately after the massage session
  Contraction time is the time between 10% and 90% of the muscle displacement after the electrical stimulation. Measuring device: TMG S2, Change = (Value after therapy - baseline)
Change in contraction time of the latissimus dorsi muscle after therapy compared to baseline. | 1) baseline, 2) immediately after the massage session
  Contraction time is the time between 10% and 90% of the muscle displacement after the electrical stimulation. Measuring device: TMG S2, Change = (Value after therapy - baseline)
Change in contraction time of the peroneus longus muscle after therapy compared to baseline. | 1) baseline, 2) immediately after the massage session
  Contraction time is the time between 10% and 90% of the muscle displacement after the electrical stimulation. Measuring device: TMG S2, Change = (Value after therapy - baseline)
Change in sustain time of the deltoid muscle after therapy compared to baseline. | 1) baseline, 2) immediately after the massage session
  Sustain time is the time between 50% of maximum contraction to 50% of maximum relaxation of a muscle after the electrical stimulation. Measuring device: TMG S2, Change = (Value after therapy - baseline)
Change in sustain time of the latissimus dorsi muscle after therapy compared to baseline. | 1) baseline, 2) immediately after the massage session
  Sustain time is the time between 50% of maximum contraction to 50% of maximum relaxation of a muscle after the electrical stimulation. Measuring device: TMG S2, Change = (Value after therapy - baseline)
Change in sustain time of the peroneus longus muscle after therapy compared to baseline. | 1) baseline, 2) immediately after the massage session
  Sustain time is the time between 50% of maximum contraction to 50% of maximum relaxation of a muscle after the electrical stimulation. Measuring device: TMG S2, Change = (Value after therapy - baseline)
Change in relaxation time of the peroneus longus muscle after therapy compared to baseline. | 1) baseline, 2) immediately after the massage session
  Relaxation time is the time between 90% of maximum contraction and 50% of maximum relaxation of a muscle after the electrical stimulation. Measuring device: TMG S2, Change = (Value after therapy - baseline)
Change in relaxation time of the deltoid muscle after therapy compared to baseline. | 1) baseline, 2) immediately after the massage session
  Relaxation time is the time between 90% of maximum contraction and 50% of maximum relaxation of a muscle after the electrical stimulation. Measuring device: TMG S2, Change = (Value after therapy - baseline)
Change in relaxation time of the latissimus dorsi muscle after therapy compared to baseline. | 1) baseline, 2) immediately after the massage session
  Relaxation time is the time between 90% of maximum contraction and 50% of maximum relaxation of a muscle after the electrical stimulation. Measuring device: TMG S2, Change = (Value after therapy - baseline)
Change in oscillation frequency of the deltoid muscle after therapy compared to baseline. | 1) baseline, 2) immediately after the massage session
  The oscillation frequency characterizes the tension of muscle tissue. Measuring device: MyotonPRO, Change = (Value after therapy - baseline)
Change in oscillation frequency of the latissimus dorsi muscle after therapy compared to baseline. | 1) baseline, 2) immediately after the massage session
  The oscillation frequency characterizes the tension of muscle tissue. Measuring device: MyotonPRO, Change = (Value after therapy - baseline)
Change in oscillation frequency of the peroneus longus muscle after therapy compared to baseline. | 1) baseline, 2) immediately after the massage session
  The oscillation frequency characterizes the tension of muscle tissue. Measuring device: MyotonPRO, Change = (Value after therapy - baseline)
Change in dynamic stiffness of the deltoid muscle muscle after therapy compared to baseline. | 1) baseline, 2) immediately after the massage session
  The dynamic stiffness corresponds to the soft tissues' capacity to resist external forces. Measuring device: MyotonPRO, Change = (Value after therapy - baseline)
Change in dynamic stiffness of the latissimus dorsi muscle after therapy compared to baseline. | 1) baseline, 2) immediately after the massage session
  The dynamic stiffness corresponds to the soft tissues' capacity to resist external forces. Measuring device: MyotonPRO, Change = (Value after therapy - baseline)
Change in dynamic stiffness of the peroneus longus muscle after therapy compared to baseline. | 1) baseline, 2) immediately after the massage session
  The dynamic stiffness corresponds to the soft tissues' capacity to resist external forces. Measuring device: MyotonPRO, Change = (Value after therapy - baseline)
Change in logarithmic decrement of the deltoid muscle after therapy compared to baseline. | 1) baseline, 2) immediately after the massage session
  Logarithmic decrement is the dissipation of the tissue oscillation. Measuring device: MyotonPRO, Change = (Value after therapy - baseline)
Change in logarithmic decrement of the latissimus dorsi muscle after therapy compared to baseline. | 1) baseline, 2) immediately after the massage session
  Logarithmic decrement is the dissipation of the tissue oscillation. Measuring device: MyotonPRO, Change = (Value after therapy - baseline)
Change in logarithmic decrement of the peroneus longus muscle after therapy compared to baseline. | 1) baseline, 2) immediately after the massage session
  Logarithmic decrement is the dissipation of the tissue oscillation. Measuring device: MyotonPRO, Change = (Value after therapy - baseline)
Change in mechanical stress relaxation time of the deltoid muscle after therapy compared to baseline. | 1) baseline, 2) immediately after the massage session
  Mechanical stress relaxation time is the time needed for the muscle to recover to its initial shape. Measuring device: MyotonPRO, Change = (Value after therapy - baseline)
Change in mechanical stress relaxation time of the latissimus dorsi muscle after therapy compared to baseline. | 1) baseline, 2) immediately after the massage session
  Mechanical stress relaxation time is the time needed for the muscle to recover to its initial shape. Measuring device: MyotonPRO, Change = (Value after therapy - baseline)
Change in mechanical stress relaxation time of the peroneus longus muscle after therapy compared to baseline. | 1) baseline, 2) immediately after the massage session
  Mechanical stress relaxation time is the time needed for the muscle to recover to its initial shape. Measuring device: MyotonPRO, Change = (Value after therapy - baseline)
Change in creep of the deltoid muscle after therapy compared to baseline. | 1) baseline, 2) immediately after the massage session
  Creep is the ratio of relaxation (R) and time between the beginning of the mechanical impulse and the time point of maximal displacement Measuring device: MyotonPRO, Change = (Value after therapy - baseline)
Change in creep of the latissimus dorsi muscle after therapy compared to baseline. | 1) baseline, 2) immediately after the massage session
  Creep is the ratio of relaxation (R) and time between the beginning of the mechanical impulse and the time point of maximal displacement Measuring device: MyotonPRO, Change = (Value after therapy - baseline)
Change in creep of the peroneus longus muscle after therapy compared to baseline. | 1) baseline, 2) immediately after the massage session
  Creep is the ratio of relaxation (R) and time between the beginning of the mechanical impulse and the time point of maximal displacement Measuring device: MyotonPRO, Change = (Value after therapy - baseline)

CONTACTS AND LOCATIONS:
Overall Officials: Marcin Piwecki, MSc, Principal Investigator — Doctoral School of Physical Culture Science, University of Physical Education in Kraków, Poland
Locations (1):
- Wroclaw University of Health and Sport Sciences, Wroclaw, Poland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bordoni B, Myers T. A Review of the Theoretical Fascial Models: Biotensegrity, Fascintegrity, and Myofascial Chains. Cureus. 2020 Feb 24;12(2):e7092. doi: 10.7759/cureus.7092. PMID 32226693
- [Background] Swanson RL 2nd. Biotensegrity: a unifying theory of biological architecture with applications to osteopathic practice, education, and research--a review and analysis. J Am Osteopath Assoc. 2013 Jan;113(1):34-52. doi: 10.7556/jaoa.2013.113.1.34. PMID 23329804